CLINICAL TRIAL: NCT05314517
Title: A Randomized, Double-blind, Placebo-Controlled Phase 2 Study With Open-label Extension to Assess the Efficacy and Safety of Namilumab in Subjects With Chronic Pulmonary Sarcoidosis
Brief Title: A Study to Assess the Efficacy and Safety of Namilumab in Participants With Chronic Pulmonary Sarcoidosis
Acronym: RESOLVE-Lung
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Kinevant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KIN-1902-2001
Record Dates: First submitted 2022-03-30; First posted 2022-04-06 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-07

CONDITIONS: Sarcoidosis, Pulmonary
MeSH Terms: conditions — Sarcoidosis, Pulmonary | interventions — namilumab

STUDY DESIGN:
Intervention Model Description: A double-blinded, randomized, placebo-controlled, parallel group design has been selected for the study. All participants, regardless of treatment assignment in the Double-blind Treatment Period, may participate in the Open Label Extension period of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug will be provided in a blinded fashion and packaged and labeled to protect the blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm 1 (Experimental): Namilumab
  Interventions: Drug: Namilumab
- Treatment Arm 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Namilumab — Namilumab administered subcutaneously
  Arms: Treatment Arm 1
Drug: Placebo — Placebo administered subcutaneously to match namilumab dosing
  Arms: Treatment Arm 2

SUMMARY:
This is a randomized, double-blind, placebo-controlled study with an open-label extension (OLE).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study with an OLE.

Participants will be randomized to receive namilumab or placebo in the 26-week Double-blind Treatment Period of the study. Namilumab, or placebo, will be administered subcutaneously (SC) every 4 weeks through Week 22 after the initial dosing period.

All participants who complete the 26-week Double-blind Treatment Period, may be eligible to participate in the 28-week OLE.

Further details are in the protocol.

ELIGIBILITY:
Inclusion Criteria :

* Male or female age ≥18 years
* Able and willing to provide written informed consent, which includes compliance with study requirements and restrictions listed in the consent form
* Greater than or equal to 6-month history of documented sarcoidosis including histological confirmation in the subject's medical records
* Evidence of sarcoidosis as indicated by: a) HRCT consistent with Pulmonary Sarcoidosis AND; b) Medical Research Council Dyspnea scale >1 (i.e., Grade 2 or more) AND; c) One or more of the following is present: i) Screening FDG-PET scan consistent with active pulmonary sarcoidosis AND SUVmax ≥ 3; ii) Recent history of worsening sarcoidosis; iii) Recent history that tapering OCS and/or ISTs resulted in an increase of pulmonary disease
* Body Mass Index (BMI) ≤ 40 kg/m2 at Screening
* Vaccinations for COVID-19 with completion of the primary series at least 2 weeks prior to randomization

Exclusion Criteria

* Hospitalized for any respiratory illness ≤ 30 days prior to or during Screening
* Greater than or equal to 20% fibrosis as indicated on HRCT-scan assessed by central read prior to randomization
* Hemoglobin ≤ 9.5 g/dL
* Participation in another interventional clinical trial (IP/Device) within 6 months prior to Screening, during screening and throughout the duration of the study
* ECG abnormalities that warrant further clinical investigation or management at Screening
* Systolic blood pressure (SBP) <90 or >180mm Hg; Diastolic blood pressure (DBP) <60 or >110 mm Hg at Screening
* Has documented laboratory-confirmed SARS-CoV-2 infection with pulmonary involvement or signs/symptoms of long COVID as determined by approved testing ≤ 6 months prior to randomization
* Other significant pulmonary disease or conditions that prevent subject from performing acceptable spirometry
* Females who are pregnant or breastfeeding or intend to be during the course of the study
* Any other acute or chronic medical condition, psychiatric condition, or laboratory abnormality, that in the judgment of the Investigator or Sponsor, may increase the risk associated with study participation or investigational product administration, or may interfere with the interpretation of study results, and would make the participant inappropriate for entry into this study
* Subjects who are treatment naive

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2025-04-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (46):
- United States (24):
  - Kinevant Study Site, Birmingham, Alabama
  - Kinevant Study Site, Palo Alto, California
  - Kinevant Study Site, Valencia, California
  - Kinevant Study Site, Denver, Colorado
  - Kinevant Study Site, Gainesville, Florida
  - Kinevant Study Site, Augusta, Georgia
  - Kinevant Study Site, Chicago, Illinois
  - Kinevant Study Site, Iowa City, Iowa
  - Kinevant Study Site, Kansas City, Kansas
  - Kinevant Study Site, New Orleans, Louisiana
  - Kinevant Study Site, Baltimore, Maryland
  - Kinevant Study Site, Minneapolis, Minnesota
  - Kinevant Study Site, Rochester, Minnesota
  - Kinevant Study Site, Greenville, North Carolina
  - Kinevant Study Site, Cincinnati, Ohio
  - Kinevant Study Site, Cleveland, Ohio
  - Kinevant Study Site, Philadelphia, Pennsylvania
  - Kinevant Study Site, Pittsburgh, Pennsylvania
  - Kinevant Study Site, Charleston, South Carolina
  - Kinevant Study Site, Rock Hill, South Carolina
  - Kinevant Study Site, Dallas, Texas
  - Kinevant Study Site, Houston, Texas
  - Kinevant Study Site, Charlottesville, Virginia
  - Kinevant Study Site, Falls Church, Virginia
- Belgium (4):
  - Kinevant Study Site, Brussels
  - Kinevant Study Site, Leuven
  - Kinevant Study Site, Liège
  - Kinevant Study Site, Yvoir
- France (3):
  - Kinevant Study Site, Bobigny
  - Kinevant Study Site, Lille
  - Kinevant Study Site, Paris
- Germany (5):
  - Kinevant Study Site, Berlin
  - Kinevant Study Site, Essen
  - Kinevant Study Site, Freiburg im Breisgau
  - Kinevant Study Site, Hanover
  - Kinevant Study Site, Heidelberg
- Netherlands (3):
  - Kinevant Study Site, Leiden
  - Kinevant Study Site, Nieuwegein
  - Kinevant Study Site, Rotterdam
- Turkey (Türkiye) (4):
  - Kinevant Study Site, Ankara
  - Kinevant Study Site, Istanbul
  - Kinevant Study Site, Izmir
  - Kinevant Study Site, Mersin
- United Kingdom (3):
  - Kinevant Study Site, Cambridge
  - Kinevant Study Site, Cottingham
  - Kinevant Study Site, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a double-blind (DB) period and an open-label extension (OLE) period.
Groups:
- Namilumab: Participants received namilumab subcutaneously (SC) on Day 1, Day 15 (Week 2), and then every 4 weeks (Q4W) thereafter through Week 22.
- Placebo: Participants received placebo matched to namilumab dosing through Week 22.
- Namilumab to Namilumab: Participants who previously received namilumab in the double-blind period received namilumab SC at week 26 and then Q4W thereafter through Week 50.
- Placebo to Namilumab: Participants who previously received placebo in the double-blind period received namilumab SC at week 26 and then Q4W thereafter through Week 50.
Period: Double-blind Period
Arm/Group | Namilumab | Placebo | Namilumab to Namilumab | Placebo to Namilumab
Started | 53 | 54 | 0 | 0
Safety Population (All randomized participants who received any amount of study treatment.) | 52 | 54 | 0 | 0
Modified Intent-to-treat (mITT) Population (All randomized participants who received any amount of DB study treatment excluding participants with a quality event.) | 49 | 51 | 0 | 0
Completed | 48 | 53 | 0 | 0
Not Completed | 5 | 1 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0 | 0
Not completed — Noncompliance | 0 | 1 | 0 | 0
Not completed — Randomized, not treated | 1 | 0 | 0 | 0
Period: Open-label Extension
Arm/Group | Namilumab | Placebo | Namilumab to Namilumab | Placebo to Namilumab
Started | 0 | 0 | 47 | 49
Safety Population | 0 | 0 | 47 | 49
Completed | 0 | 0 | 30 | 29
Not Completed | 0 | 0 | 17 | 20
Not completed — Adverse Event | 0 | 0 | 1 | 2
Not completed — Investigator decision | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2
Not completed — Use of prohibited medication | 0 | 0 | 1 | 0
Not completed — Sponsor decision to terminate study | 0 | 0 | 13 | 15

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who receive any amount of study treatment.
Groups:
- Namilumab: Participants received namilumab SC on Day 1, Day 15 (Week 2), and then Q4W thereafter through Week 22.
- Total: Total of all reporting groups
Arm/Group | Namilumab | Placebo | Total
Number analyzed (Participants) | 52 | 54 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (12.13) | 54.1 (10.35) | 52.9 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 29 | 32 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 50 | 49 | 99
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 43 | 45 | 88
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Rescue Event During the DB Period
Description: Rescue events included: Participants with worsening sarcoidosis requiring rescue treatment; and participants failing to follow protocol defined concomitant sarcoidosis medication requirements (oral corticosteroids [OCS] taper/immunosuppressive therapy [IST] removal/prohibited medication). Participants with premature treatment discontinuation in the DB period without rescue event were considered as with missing rescue event status and excluded from analysis.
Time Frame: Baseline to Week 26 for participants continuing to OLE and up to Week 30 for participants not continuing to OLE, as rescue events occurring within 8 weeks of last dose were included in the analysis for participants not continuing to the OLE period.
Population: mITT population included all randomized participants who received any amount of DB study treatment, excluding participants with a quality event. 'Overall number of participants analyzed' = participants with rescue event status.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Namilumab | Placebo
Number analyzed (Participants) | 48 | 51
percentage of participants | 37.5 [27.0 to 49.4] | 23.5 [15.2 to 34.5]
Statistical Analysis 1: Comparison: Namilumab vs Placebo; Test type: Other; p = 0.1244, Cochran-Mantel-Haenszel; Stratified Common Risk Difference = 14.1, 90% CI 2-sided [-1.0 to 29.2]

2. Secondary Outcome: Change From Baseline in Percent Predicted Forced Vital Capacity (FVC) at Week 26
Description: FVC is the volume of air (in liters) that can be forcibly blown out after full inspiration in the upright position. Percent of predicted FVC = (actual FVC measurement)/(predicted value of FVC) * 100. Least square (LS) mean and standard error (SE) were calculated using mixed model for repeated measure (MMRM).
Time Frame: Baseline, Week 26
Population: The mITT population included all randomized participants who received any amount of DB study treatment, excluding participants with a quality event. 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted FVC
Arm/Group | Namilumab | Placebo
Number analyzed (Participants) | 49 | 51
percentage of predicted FVC | -3.28 (1.058) | -2.92 (0.967)

3. Secondary Outcome: Time to the First Rescue Event During the DB Period
Description: Time of first rescue event was defined as the time from randomization to the rescue event date. Rescue events included: Participants with worsening sarcoidosis requiring rescue treatment; and participants failing to follow protocol defined concomitant sarcoidosis medication requirements (OCS taper/IST removal/prohibited medication). Data was calculated using the Kaplan-Meier estimator.
Time Frame: as for outcome 1
Population: mITT population included all randomized participants who received any amount of DB study treatment, excluding participants with a quality event.
Measure: Median (Full Range); unit: weeks
Arm/Group | Namilumab | Placebo
Number analyzed (Participants) | 49 | 51
weeks | 11.0 [1.0 to 26.6] | 12.86 [3.0 to 22.1]

4. Secondary Outcome: Percentage of Participants Successfully Achieving OCS Taper Without Rescue Event During the DB Period
Description: Percentage of participants achieving OCS taper (achieving OCS dose ≤5 milligrams [mg] at end of Week 10 [Day 77] for participants with baseline OCS >10 mg/day, achieving ≤ 5 mg at end of Week 6 [Day 49] for participants with baseline OCS >5 to ≤10 mg/day) without any rescue event during the DB period for participants with OCS >5 mg/day at baseline are reported.
Time Frame: Baseline to Week 26
Population: The mITT population included all randomized participants who received any amount of DB study treatment, excluding participants with a quality event. 'Overall number of participants analyzed' = participants with OCS >5 mg/day at baseline.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Namilumab | Placebo
Number analyzed (Participants) | 15 | 13
percentage of participants | 53.3 [33.3 to 72.3] | 76.9 [54.2 to 90.4]

5. Secondary Outcome: Change From Baseline in the Kings Sarcoidosis Questionnaire (KSQ) Lung Domain Score at Week 26
Description: The KSQ has 29 questions (items 1 to 16, and items 26-38). The KSQ Lung domain score was calculated based on items 11 to 16. Each item was answered on a 7-point scale where 1 means the participant experienced symptoms all the time and 7 means the participant did not experience the symptom at all. The raw item scores were first converted into item re-scores using the first conversion step. Then, the re-scores for the 6 items were totaled and the total converted into the logit 1 (worst symptom) - 100 (no symptom) score, where higher score indicating better health. LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Namilumab | Placebo
Number analyzed (Participants) | 47 | 49
units on a scale | 1.61 (1.866) | 3.47 (1.771)

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) During the DB Period
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered the study drug and which did not necessarily have a causal relationship with this treatment. TEAEs are those AEs with start date on or after the start date of treatment through the earlier of 18-week post last dose during DB period or prior to first dose during OLE period, whichever was earlier. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Baseline up to Week 26
Population: Safety population included all randomized participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Namilumab | Placebo
Number analyzed (Participants) | 52 | 54
Participants | 49 | 51

ADVERSE EVENTS:
Time Frame: From first dose to 18 weeks after last dose (up to 68 weeks)
Description: Safety population included all randomized participants who received any amount of study treatment. Per protocol, the Safety on-namilumab population (namilumab to namilumab) included all randomized participants who received any amount of namilumab during the DB or OLE period. Each arm includes all AEs in randomized participants from first dose of namilumab in DB or OLE period until 18 weeks after last dose.
Groups:
- Namilumab to Namilumab: Participants received namilumab SC on Day 1, Day 15 (Week 2), and then Q4W thereafter through Week 22.
  Participants then received namilumab SC at week 26 and then Q4W thereafter through Week 50.
Arm/Group | Namilumab | Placebo | Namilumab to Namilumab | Placebo to Namilumab
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/54 | 0/52 | 0/49
Serious Adverse Events (participants affected / at risk) | 3/52 | 3/54 | 7/52 | 5/49
Other Adverse Events (participants affected / at risk) | 49/52 | 51/54 | 51/52 | 44/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Namilumab (N=52) | Placebo (N=54) | Namilumab to Namilumab (N=52) | Placebo to Namilumab (N=49)
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Conduction disorder (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Namilumab (N=52) | Placebo (N=54) | Namilumab to Namilumab (N=52) | Placebo to Namilumab (N=49)
Upper respiratory tract infection (Infections and infestations) | 5 | 11 | 12 | 10
Nasopharyngitis (Infections and infestations) | 6 | 3 | 9 | 2
Bronchitis (Infections and infestations) | 2 | 4 | 3 | 3
Influenza (Infections and infestations) | 3 | 3 | 4 | 3
Urinary tract infection (Infections and infestations) | 3 | 3 | 5 | 1
COVID-19 (Infections and infestations) | 3 | 2 | 6 | 2
Sinusitis (Infections and infestations) | 0 | 3 | 2 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 1
Rhinitis (Infections and infestations) | 1 | 1 | 1 | 1
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Borrelia infection (Infections and infestations) | 1 | 0 | 1 | 0
Bronchitis haemophilus (Infections and infestations) | 1 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 2 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 2 | 0
Gastrointestinal bacterial infection (Infections and infestations) | 1 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 1 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Pericoronitis (Infections and infestations) | 1 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Post-acute COVID-19 syndrome (Infections and infestations) | 1 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 1
Tinea versicolour (Infections and infestations) | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 1 | 1
Viral infection (Infections and infestations) | 1 | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 3 | 0 | 3 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Monocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 2 | 0 | 2 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 1 | 1
Sarcoidosis (Immune system disorders) | 0 | 1 | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 1 | 1
Sleep disorder (Psychiatric disorders) | 1 | 1 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 4
Mood altered (Psychiatric disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 4 | 4 | 5
Dizziness (Nervous system disorders) | 4 | 1 | 6 | 1
Dysgeusia (Nervous system disorders) | 2 | 1 | 2 | 0
Essential tremor (Nervous system disorders) | 1 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1 | 0
Migraine with aura (Nervous system disorders) | 0 | 1 | 0 | 0
Ophthalmic migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 1 | 0
Small fibre neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 2 | 0 | 2 | 0
Visual impairment (Eye disorders) | 2 | 0 | 2 | 0
Conjunctival deposit (Eye disorders) | 1 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 1 | 0
Hypermetropia (Eye disorders) | 0 | 1 | 0 | 0
Macular degeneration (Eye disorders) | 1 | 0 | 1 | 0
Meibomian gland dysfunction (Eye disorders) | 0 | 1 | 0 | 0
Myopia (Eye disorders) | 1 | 0 | 1 | 0
Photophobia (Eye disorders) | 1 | 0 | 2 | 0
Retinal tear (Eye disorders) | 0 | 1 | 0 | 0
Swelling of eyelid (Eye disorders) | 1 | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 1 | 0
Visual field defect (Eye disorders) | 1 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1 | 2 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac sarcoidosis (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 2 | 2
Hypertensive urgency (Vascular disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 15 | 19 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 10 | 12 | 5
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 13 | 16
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 6 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Larynx irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung hyperinflation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 4 | 6 | 3
Constipation (Gastrointestinal disorders) | 3 | 4 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 7 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 4 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Liver sarcoidosis (Hepatobiliary disorders) | 1 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 4 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Cutaneous sarcoidosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Ephelides (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 4 | 12 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 4 | 5 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 6 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/29 | 0/32 | 1/29 | 0/29 — This is a sex-specific AE. Only male participants were at risk.
Dyspareunia (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 10 | 6 | 12 | 5
Injection site pain (General disorders) | 5 | 3 | 5 | 0
Non-cardiac chest pain (General disorders) | 4 | 2 | 4 | 0
Oedema peripheral (General disorders) | 0 | 3 | 0 | 1
Chest discomfort (General disorders) | 0 | 3 | 0 | 1
Chills (General disorders) | 0 | 3 | 1 | 0
Injection site reaction (General disorders) | 1 | 2 | 1 | 1
Injection site erythema (General disorders) | 1 | 1 | 1 | 1
Asthenia (General disorders) | 2 | 0 | 4 | 0
Injection site haematoma (General disorders) | 2 | 0 | 2 | 0
Pain (General disorders) | 1 | 1 | 3 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 3 | 5
Injection site rash (General disorders) | 1 | 0 | 1 | 0
Facial pain (General disorders) | 1 | 0 | 1 | 1
Feeling hot (General disorders) | 0 | 1 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 1 | 0
Injection site paraesthesia (General disorders) | 1 | 0 | 1 | 0
Injection site pruritus (General disorders) | 1 | 0 | 1 | 0
Injection site swelling (General disorders) | 0 | 1 | 0 | 0
Injection site warmth (General disorders) | 0 | 1 | 0 | 0
Injury associated with device (General disorders) | 1 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 1 | 2 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 3 | 1
Hepatic enzyme increased (Investigations) | 1 | 1 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 1 | 2 | 0
Surfactant protein increased (Investigations) | 2 | 0 | 3 | 1
Weight decreased (Investigations) | 1 | 1 | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 4 | 1
Blood glucose increased (Investigations) | 1 | 0 | 2 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 1 | 0
Eosinophil count increased (Investigations) | 1 | 0 | 2 | 1
Forced vital capacity decreased (Investigations) | 1 | 0 | 1 | 1
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 1 | 0
Haematocrit increased (Investigations) | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 1 | 0
High density lipoprotein increased (Investigations) | 1 | 0 | 1 | 0
Hysteroscopy (Investigations) | 1 | 0 | 1 | 0
Influenza A virus test positive (Investigations) | 1 | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 1 | 0 | 1 | 0
Lung diffusion test decreased (Investigations) | 0 | 1 | 0 | 1
Pulmonary function test decreased (Investigations) | 0 | 1 | 0 | 0
Stool analysis (Investigations) | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 3 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Complications of transplanted lung (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Environmental exposure (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Tattoo associated skin reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Gingival recession (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Crystal urine present (Investigations) | 1 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 1
Hepatitis E (Infections and infestations) | 0 | 0 | 0 | 1
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 0 | 1 | 0
Norovirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Emotional poverty (Psychiatric disorders) | 0 | 0 | 0 | 1
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 1 | 0
Dementia (Nervous system disorders) | 0 | 0 | 1 | 0
Hyposmia (Nervous system disorders) | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Sedation (Nervous system disorders) | 0 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Childhood asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Granulomatous liver disease (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Shoulder girdle pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Porokeratosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Vaccination site pain (General disorders) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 2
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 1 | 0
Bacterial test positive (Investigations) | 0 | 0 | 1 | 0
Band neutrophil count increased (Investigations) | 0 | 0 | 1 | 0
Blood bicarbonate increased (Investigations) | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0
Blood creatine increased (Investigations) | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1
Full blood count decreased (Investigations) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Lymphocyte morphology abnormal (Investigations) | 0 | 0 | 1 | 0
Oxygen consumption increased (Investigations) | 0 | 0 | 1 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 1
Pulmonary function test abnormal (Investigations) | 0 | 0 | 0 | 1
Pulmonary function test increased (Investigations) | 0 | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural headache (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT05314517/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT05314517/SAP_001.pdf